CLINICAL TRIAL: NCT01716923
Title: A Randomized Controlled Double-Blind Phase 3 Study to Assess Characteristics of S 303 Treated RBC Components and Evaluate Safety and Efficacy in Patients Requiring Transfusion Support of Acute Anemia
Brief Title: Study to Assess S303 RBCs and Evaluate Safety and Efficacy in Patients Requiring Transfusion Support of Acute Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cerus Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: CLI 00070
Record Dates: First submitted 2012-10-26; First posted 2012-10-30 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-06

CONDITIONS: Focus:Use of S303 RBCs in Patients With Acute Anemia
MeSH Terms: interventions — Erythrocyte Count; Congresses as Topic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- S-303 Treated Red Blood Cells (Experimental): Patients receive S-303 treated red blood cells (RBCs).
  Interventions: Biological: S-303 Red Blood Cells (RBCs) - Test
- Conventional, untreated Red Blood Cells (Active Comparator): Patients receive conventional, untreated red blood cells (RBCs).
  Interventions: Biological: Conventional, untreated red blood cells (RBCs) - Control

INTERVENTIONS:
Biological: S-303 Red Blood Cells (RBCs) - Test
  Arms: S-303 Treated Red Blood Cells
Biological: Conventional, untreated red blood cells (RBCs) - Control
  Arms: Conventional, untreated Red Blood Cells

SUMMARY:
The clinical study will assess the in-vitro characteristics of red blood cells (RBCs) per the European Union (EU) criteria for leukocyte depleted RBCs in additive solution and evaluate the safety and efficacy of S-303 treated RBCs in a patient population requiring RBC transfusion support for acute anemia.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, of either gender.
2. Must be willing to use an acceptable form of contraceptive while on study (as approved by the Investigator or designee)
3. Must be readily available by telephone
4. Must provide an informed consent for study participation and have signed an ethics committee (EC)-approved informed consent
5. Must have a negative cross match to S 303 red blood cells (RBCs) at study entry
6. Must have a blood type of either A+ or O+
7. Patients must have a likelihood of receiving a transfusion as determined by the Investigator OR a Transfusion Risk Understanding Screening Tool (TRUST) Score of ≥3 at study entry
8. Must be scheduled to receive one of the following operative procedures:

   * Coronary artery bypass graft only, first procedure
   * Valve repair or replacement only, first procedure
   * A combination of first time Coronary Artery Bypass Graft (CABG) and valve repair or replacement

After consultation with the Medical Monitor, provision can be made to enroll patients who may meet these general criteria but whose surgical procedure is not precisely described in the above categories. Such patients will be classified as "other" with their explicit condition reported with other study data.

Exclusion Criteria:

1. A positive pregnancy test result
2. Inability of patient to comply with the protocol in the opinion of the Investigator or attending physician
3. Breast-feeding of an infant or child
4. Active autoimmune hemolytic anemia, or a positive Direct Antiglobulin Test (DAT) result
5. Treatment with any medication that is known to adversely affect red blood cell viability
6. Emergent or salvage surgical status at the time of surgery defined as follows:

   * Presence of ongoing ischemia including angina at rest despite maximal medical therapy
   * Acute evolving myocardial infarction within 24 hours before surgery
   * Pulmonary edema requiring intubation
   * Presence of shock or hemodynamic instability with or without circulatory support
   * Systolic blood pressure < 80 mm Hg and/or Cardiac Index < 1.8 despite medical intervention (intravenous inotropes or similar pharmacologic agents)
   * Cardiopulmonary resuscitation in the 24 hours prior to surgery or anesthesia induction
   * Requiring an intra-aortic balloon pump or ventricular assist device
7. Participation in any one of the following types of clinical studies either concurrently or within the previous 28 days: investigational blood products, pharmacologic agents or imaging materials, including dyes, investigational surgical techniques, or devices. Studies of nutrition, psychology, or socioeconomic issues are not grounds for exclusion
8. Current diagnosis of either chronic or acute renal failure (requiring dialysis) or a serum creatinine greater than or equal to 1.8 mg/dL within 30 days prior to the start of surgery
9. Current diagnosis of either chronic or acute hepatic insufficiency or a total serum bilirubin greater than or equal to 2.0 mg/dL within 30 days prior to the start of surgery
10. Pre-existing RBC antibody that may make the provision of compatible study red blood cell (RBC) components difficult
11. Patients requiring plasma removal or irradiation of the RBC
12. Patients with prior history of severe allergic transfusion reactions
13. A positive cross match to S 303 treated RBC

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-04; Primary Completion 2014-07 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint - mean hemoglobin content | Day 2
  The mean hemoglobin content per red blood cell (RBC) component compared between the treatment groups
Primary Safety Endpoint - Adverse events | 90 days
  The frequency of adverse events (related and unrelated to study RBC components) will be compared between the treatment groups.

SECONDARY OUTCOMES:
Secondary Efficacy Endpoint | Day 35
  Proportion of RBC components that have adenosine-5'-triphosphate (ATP) levels of greater than 2 μmol/L
Secondary Efficacy Endpoint | Day 35
  Proportion of RBC components that meet the European Union (EU) guideline for hemoglobin content, hematocrit, and hemolysis at the end of storage
Secondary Efficacy Endpoint | Day 35
  Proportion of RBC components that have plasma-free hemoglobin levels corresponding to ≤ 0.8% hemolysis

OTHER OUTCOMES:
Exploratory Endpoint - incidence of renal insufficiency | Daily on days 0 through 6
  Incidence of renal insufficiency, indicated by serum creatinine level >2 mg/dL WITH at least a 50% increase from pre-operative baseline OR a new requirement for therapy to treat renal insufficiency (dialysis)
Exploratory Endpoint - incidence of hepatic insufficiency | Daily on days 0 through 6
  Incidence of hepatic insufficiency, indicated by total bilirubin that is >2 times the upper limit of normal AND represents at least a 50% increase from the preoperative baseline
Exploratory endpoint - Cardiopulmonary function | Day 7 and 13
  Cardiopulmonary function at the time of first ambulation and at the time of discharge, as measured by a standardized 6 Minute Walk Test (6MWT)

CONTACTS AND LOCATIONS:
Overall Officials: Arndt H Kiessling, MD, Principal Investigator — Klinikum der J.-W.-G.-Universität Frankfurt; Katharina Madlener, Dr, Principal Investigator — Kerckhoff-Klinic GmbH
Locations (2):
- Germany (2):
  - Kerckhoff-Klinic GmbH, Bad Nauheim, Hesse
  - Klinikum der J.-W.-G.-Universität Frankfurt, Frankfurt

REFERENCES:
- [Derived] Brixner V, Kiessling AH, Madlener K, Muller MM, Leibacher J, Dombos S, Weber I, Pfeiffer HU, Geisen C, Schmidt M, Henschler R, North A, Huang N, Mufti N, Erickson A, Ernst C, Rico S, Benjamin RJ, Corash LM, Seifried E. Red blood cells treated with the amustaline (S-303) pathogen reduction system: a transfusion study in cardiac surgery. Transfusion. 2018 Apr;58(4):905-916. doi: 10.1111/trf.14528. Epub 2018 Mar 1. PMID 29498049